CLINICAL TRIAL: NCT03656263
Title: The Clinical Significance of Portal Hypertension After Cardiac Surgery
Brief Title: The Clinical Significance of Portal Hypertension After Cardiac Surgery: a Multicenter Prospective Observational Study
Acronym: TECHNO-MULTI
Status: Completed | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Responsible Party: Principal Investigator, Andre Denault, Principal investigator, Montreal Heart Institute
Other Study IDs: TECHNO-MULTI
Record Dates: First submitted 2018-08-29; First posted 2018-09-04 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Surgery--Complications; Congestive Heart Failure; Right Heart Failure; Anesthesia; Venous Congestion
Keywords: echocardiography; Portal Doppler; Cardiac surgery
MeSH Terms: conditions — Heart Failure; Hyperemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- High risk cardiac surgery patients: Defined as either:
  * Multiple surgical procedures planned and/or,
  * EuroSCORE ≥ 5% and/or,
  * Known pulmonary hypertension (mPAP>25 mmHg or sPAP > 40 mmHg)
  Interventions: Diagnostic Test: Doppler assessment of portal vein flow

INTERVENTIONS:
Diagnostic Test: Doppler assessment of portal vein flow — Doppler assessment of portal vein flow using peri-operative trans-esophageal echography before and after cardiopulmonary bypass.

SUMMARY:
Portal flow pulsatility detected by Doppler ultrasound is an echographic marker of cardiogenic portal hypertension from right ventricular failure and is associated with adverse outcomes based on previous studies performed at the Montreal Heart Institute. This multicenter prospective cohort study aims to determine if portal flow pulsatility after cardiopulmonary bypass separation is associated with a longer requirement of life support after cardiac surgery.

DETAILED DESCRIPTION:
Hypothesis: Portal flow pulsatility detected by Doppler ultrasound during cardiac surgery is an echographic marker of cardiogenic portal hypertension from right ventricular failure and is associated with adverse clinical outcomes.

Background: Peri-operative right ventricular failure is associated with a high mortality rate. In this context, organ perfusion is hampered by both the reduction of cardiac output and venous congestion from the elevation of central venous pressure. The clinician's objective is to appreciate the hemodynamic impact on end-organs in an effort to adjust the therapy accordingly since the ultimate goal is to optimize their perfusion. Based on this rationale, organ specific blood flow assessment using Doppler ultrasound could be used to personalize management. In order to non-invasively assess the presence of cardiogenic portal hypertension, Doppler ultrasound can be used to detect portal flow pulsatility, an abnormal variation in the velocity of blood flow within the main portal vein. In two single-center cohort studies, the presence of portal flow pulsatility after cardiac surgery was independently associated with post-operative complications such as major bleeding, acute kidney injury (AKI) and delirium as well as increased length of intensive care unit (ICU) stay.

Specific Objectives: This multi-center cohort study aim to determine whether the association between portal flow pulsatility and organ dysfunction seen in previous studies is present across multiple cardiac surgery centers.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old) and able to give informed consent undergoing cardiac surgery with the use of CPB for whom peri-operative TEE is planned.
* High surgical risk defined as at least one of the following:

  1. Multiple surgical procedures planned
  2. EuroSCORE II ≥ 5%
  3. Known pulmonary hypertension (mPAP>25mmHg or sPAP>40mmHg).

Exclusion Criteria:

* Patient with a critical pre-operative state defined as vasopressor requirement, mechanical circulatory support, dialysis, mechanical ventilation or cardiac arrest necessitating resuscitation.
* Patient with known condition that could interfere with portal flow assessment or interpretation (liver cirrhosis, portal vein thrombosis)
* Planned cardiac transplantation
* Planned ventricular assist device implantation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery at high risk for complications.
Sampling Method: Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2021-02-20 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Duration of invasive life support after cardiac surgery. (Tpod) | Up to 28 days
  Defined as the time of Persistent Organ Dysfunction (POD) or Death

SECONDARY OUTCOMES:
All cause death | Up to 28 days
  Death from any cause
Acute kidney injury according to KDIGO serum creatinine criteria | Up to 28 days
  Stage 1: ≥50% or 27 umol/L increases in serum creatinine Stage 2: ≥100% increase in serum creatinine Stage 3 ≥200% increase in serum creatinine or an increase to a level of ≥254 umol/L or dialysis initiation.
Major bleeding defined by the Bleeding Academic Research Consortium (BARC) | Up to 28 days
  Perioperative intracranial bleeding within 48h Reoperation after closure of sternotomy for the purpose of controlling bleeding Transfusion of ≥5 units of whole blood of packed red blood cells within a 48 hours period Chest tube output ≥2L within a 24 hours period
Surgical reintervention for any reasons | Up to 28 days
  Re-operation after the initial surgery for any cause
Deep sternal wound infection or mediastinitis | Up to 28 days
  Diagnosis of a deep incisional surgical site infection or mediastinitis by a surgeon or attending physician.
Delirium | Up to 28 days
  Defined as a intensive care delirium screening checklist (ICDSC) score of ≥4 in the week following surgery or positive result for the Confusion Assessment Method for the ICU (CAM-ICU)
Stroke | Up to 28 days
  A central neurologic deficit persisting longer than 72 hours
Total duration of ICU stay in hours | Up to 28 days
  Number of hours passed in the ICU
Duration of hospital stay (in days) | Up to 28 days
  Number of days hospitalized from the day of surgery to discharge
Duration of mechanical ventilation (in hours) | Up to 28 days
  Number of hours of mechanical ventilation
A composite outcome of major morbidity or mortality (41): including death, prolonged ventilation, stroke, renal failure (Stage ≥2), deep sternal wound infection and reoperation for any reason. | Up to 28 days
  Composite endpoint after cardiac proposed by the Society of Thoracic Surgeons

CONTACTS AND LOCATIONS:
Overall Officials: André Denault, MD PhD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Denault A, Couture EJ, De Medicis E, Shim JK, Mazzeffi M, Henderson RA, Langevin S, Dhawan R, Michaud M, Guensch DP, Berger D, Erb JM, Gebhard CE, Royse C, Levy D, Lamarche Y, Dagenais F, Deschamps A, Desjardins G, Beaubien-Souligny W. Perioperative Doppler ultrasound assessment of portal vein flow pulsatility in high-risk cardiac surgery patients: a multicentre prospective cohort study. Br J Anaesth. 2022 Nov;129(5):659-669. doi: 10.1016/j.bja.2022.07.053. Epub 2022 Sep 30. PMID 36184294